CLINICAL TRIAL: NCT02862652
Title: Role of the Microparticles and of Tissue Factor in the Pro-thrombotic Phenotype and the Thromboembolic Complications During the Acute Lymphoblastic Leukemia in Children
Acronym: THROMBLEUKEMIA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CHU de Reims (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: PA13047
Record Dates: First submitted 2016-08-08; First posted 2016-08-11 (Estimated); Last update posted 2026-01-21 (Actual); Status verified 2017-03

CONDITIONS: Acute Lymphoblastic Leukemia
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Blood Specimen Collection

ARMS (1):
- children with acute lymphoblastic leukemia (Experimental)
  Interventions: Other: Blood sample

INTERVENTIONS:
Other: Blood sample — Blood sample to quantify microparticles and to study expression and activity of the tissue factor on their surface

SUMMARY:
Acute lymphoblastic leukemia is the most common malignancy of the child. Current therapeutic strategies allow healing of over 80% of children. However these treatments are associated with toxicity, with a mortality of 1-2%. The most frequent complications, occuring during treatment initiation, are the thromboembolic complications.

The most commonly accepted explanation is that of an anti-thrombin depletion by chemotherapy used in the treatment, L-asparaginase. But the anti-thrombin supplementation showed no efficacy in the prevention of these thromboembolic complications. Therefore most authors consider that a multifactorial mechanism is behind these events, involving both treatment and malignant cells. The interaction of these two factors participate in the damage of the vascular endothelium.

The microparticles are membrane fragments derived from budding from the membrane of activated cells or apoptosis. Their thrombogenic role is linked to the expression of coagulation activators such as tissue factor. It is also associated with their role in the modulation of signaling pathways involved in the invasiveness and angiogenesis in endothelial cells.

In acute lymphoblastic leukemia, the presence and role of microparticles have not been studied. Our hypothesis is that of production of microparticles upon lysis of blasts then upon activation of endothelial cells induced by the induction therapy, participating in a procoagulant phenotype.

DETAILED DESCRIPTION:
The aims of this study are

* quantify the microparticles in children receiving induction therapy for Acute lymphoblastic leukemia at diagnosis and during treatment
* study the origin of these particles and the expression and activity of the tissue factor on their surface, at diagnosis and during treatment

ELIGIBILITY:
Inclusion Criteria:

* children with acute lymphoblastic leukemia
* children and their parents consenting to participate to the study
* children enrolled in the national healthcare insurance program

Max Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 24 (Actual)
Dates: Start 2014-05 (Actual); Primary Completion 2017-03-21 (Actual); Study Completion 2017-03-21 (Actual)

PRIMARY OUTCOMES:
Presence of microparticules | Day 0
  Presence of microparticles investigated using flow cytometry

SECONDARY OUTCOMES:
Presence of microparticules | Day 8
  Presence of microparticles investigated using flow cytometry
Presence of microparticules | Day 15
  Presence of microparticles investigated using flow cytometry
Presence of microparticules | Day 25
  Presence of microparticles investigated using flow cytometry
Presence of microparticules | Day 36
  Presence of microparticles investigated using flow cytometry
expression of the tissue factor | Day 0
  expression of the tissue factor investigated using flow cytometry
expression of the tissue factor | Day 3
  expression of the tissue factor investigated using flow cytometry
expression of the tissue factor | Day 15
  expression of the tissue factor investigated using flow cytometry
expression of the tissue factor | Day 25
  expression of the tissue factor investigated using flow cytometry
expression of the tissue factor | Day 36
  expression of the tissue factor investigated using flow cytometry
Thromboembolic complication | Day 36
  complication thromboembolic diagnosed by the clinical examination and by the imaging

CONTACTS AND LOCATIONS:
Locations (1):
- Chu de Reims, Reims, France

REFERENCES:
- [Background] Pluchart C, Barbe C, Poitevin G, Audonnet S, Nguyen P. A pilot study of procoagulant platelet extracellular vesicles and P-selectin increase during induction treatment in acute lymphoblastic leukaemia paediatric patients: two new biomarkers of thrombogenic risk? J Thromb Thrombolysis. 2021 Apr;51(3):711-719. doi: 10.1007/s11239-020-02346-7. Epub 2020 Nov 28. PMID 33247807